CLINICAL TRIAL: NCT06525558
Title: The Presence of Microplastics and Nanoplastics in the Humans Ileum, Colon, and Rectum and Their Relation With Inflammatory Bowel Disease (IBD): A Cross-sectional Observational Study
Brief Title: The Presence of Microplastics and Nanoplastics in the Humans Ileum, Colon, and Rectum and Their Relation With Inflammatory Bowel Disease (IBD)
Acronym: MATISSE
Status: Not yet recruiting | Type: Observational
Sponsor: Pierpaolo Sileri (Other)
Responsible Party: Sponsor-Investigator, Pierpaolo Sileri, Professor, IRCCS Ospedale San Raffaele
Organization: IRCCS Ospedale San Raffaele (Other)
Other Study IDs: MATISSE
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-10

CONDITIONS: IBD
Keywords: Microplastics; Nanoplastics; Human Intestine; IBD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — This study does not add additional risks to patients since the intestinal resection is done during surgery according to standard clinical practice. The study sample will then be collected from the resected specimen and sent to the laboratory for proper storage and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IBD Group: Patients with IBD disease (Crohn disease and Ulcerative Colitis) who will be subjected, as established by normal clinical practice, to any type of bowel surgery that involves resection of colon, ileum and/or rectum
  Interventions: Procedure: Intestinal resection
- Non-IBD Group: Patients with other diseases that are not IBD (for example, tumor, rectal prolapse or diverticulitis) who will be subjected, as established by normal clinical practice, to any type of bowel surgery that involves resection of colon, ileum and/or rectum
  Interventions: Procedure: Intestinal resection

INTERVENTIONS:
Procedure: Intestinal resection — This study does not add additional risks for patients as the resected specimen is collected during the surgery in accordance with standard clinical practice.

SUMMARY:
Based on recent studies it is hypothesized that microplastics and nanoplastics (MNPs) are present in human's ileum, colon, and rectum and that their presence may have a correlation with Inflammatory Bowel Disease (IBD).

This study is a cross-sectional, single-center, non-profit observational study. The main objectives are to define in vitro the presence of MNPs in the humans ileum, colon, and rectum and to evaluate if there is a correlation between this presence and IBD. In vitro metabolomics and proteomics analyses of the study sample and the assessment of participants' daily plastic exposure are considered exploratory objectives. For this purpose, a total of 102 patients undergoing a surgery where intestinal resection is included, will be enrolled.

DETAILED DESCRIPTION:
Based on recent studies, it is hypothesized that MNPs are present in the human's ileum, colon, and rectum and that this presence may have a correlation with Inflammatory Bowel Disease (IBD).

This study is a cross-sectional, single-center, non-profit, observational study in which filling out, una-tantum, the daily plastic exposure 10-minute questionnaire is the only additional procedure. Adult patients who will be subjected, as established by normal clinical practice, to any type of bowel surgery that involves resection of colon, ileum and/or rectum, will be included (n=102). Participants will be divided in two groups, Group IBD (n=51) and Group Non IBD (n=102).

This study does not add additional clinical practices or controls to the participants and there are not follow up visits programmed. Furthermore, this study does not add additional risks to patients since the intestinal resection is done during surgery according to standard clinical practice.

The study population includes patients who will be subjected, as established by normal clinical practice, to any type of bowel surgery that involves resection of colon, ileum and/or rectum and the study object is to determine the presence, composition, and potential health implications of microplastics and nanoplastics in the human ileum, colon, and rectum. Focusing on whether the presence of these particles correlates with intestinal inflammatory processes.

For this purpose, the primary objective of this study is to determine the presence of microplastics and nanoplastics in the humans ileum, colon, and rectum. The secondary objective is to evaluate if there is correlation between the presence of the microplastics and nanoplastics in the humans bowel and Inflammatory Bowel Disease (IBD). Finally, the exploratory objectives are to analyze further characteristics of the study sample such as the metabolomics and proteomics characteristics and to assess participants' daily plastic exposure.

The study will have a total duration of 15 months and includes 9 months of enrollment and 6 months for laboratory analysis. All the collected samples will be analyzed in vitro by the following methods:

* MNPs presence determination and characterization
* Metabolomics
* Proteomics

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo any type of bowel surgery due to any type of clinical condition, as established by normal clinical practice, where colon, ileum and/or rectum resection is involved.
* Patients aged ≥ 18 years.
* Patients who have read, understood, accepted, and signed the informed consent to the study.
* Female patients within and outside of childbearing age (breastfeeding women can be included in the study)

Exclusion Criteria:

* Patients aged < 18 years.
* Pregnant women.
* Patients who have not accepted informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients who will be subjected, as established by normal clinical practice, to any type of bowel surgery that involves resection of colon, ileum and/or rectum. The participants will be male and female subjects, with age ≥ 18 years.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Determination of the presence of microplastics and nanoplastics in the humans ileum, colon, and rectum. | Baseline/Time zero
  The variables for evaluating the primary objective:
  - Monomer Type and characterization:
  * Type
  * Concentration

SECONDARY OUTCOMES:
Evaluation of the possible correlation between the presence of the microplastics and nanoplastics in the humans bowel and Inflammatory Bowel Disease (IBD). | Baseline/Time zero
  To determine this correlation, the participants will be divided in two groups:
  1. IBD Group: Participants with IBD
     * Crohn disease (n=26)
     * Ulcerative Colitis (n=25)
  2. Non IBD Group: Participants with other diseases that are not IBD (for example, tumor, rectal prolapse or diverticulitis)
  The data collected from the two groups will be compared and evaluated using appropriate statistical methods.

OTHER OUTCOMES:
Analysis of further characteristics of the study sample such as the metabolomics and proteomics characteristics and assessment of participants' daily plastic exposure. | Baseline/Time zero
  Since the presence of MNPs might influence the primary metabolomic pathways and lead to modifications in the proteomic profiling of tissues, metabolomics and proteomics analyses will be performed to comprehensively assess any possible alteration resulting from the presence of these particles.
  Furthermore, participants' daily plastic exposure will be assessed through the 10-minute questionnarie questions defined in the "Baseline Questionary" supporting document, related to their dietary habits.

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Sileri, Prof., Principal Investigator — IRCCS Ospedale San Raffaele

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu L, Kang Y, Ma M, Wu Z, Zhang L, Hu R, Xu Q, Zhu J, Gu X, An L. Tissue accumulation of microplastics and potential health risks in human. Sci Total Environ. 2024 Mar 10;915:170004. doi: 10.1016/j.scitotenv.2024.170004. Epub 2024 Jan 12. PMID 38220018
- [Background] Ibrahim YS, Tuan Anuar S, Azmi AA, Wan Mohd Khalik WMA, Lehata S, Hamzah SR, Ismail D, Ma ZF, Dzulkarnaen A, Zakaria Z, Mustaffa N, Tuan Sharif SE, Lee YY. Detection of microplastics in human colectomy specimens. JGH Open. 2020 Nov 21;5(1):116-121. doi: 10.1002/jgh3.12457. eCollection 2021 Jan. PMID 33490620
- [Background] Yan Z, Liu Y, Zhang T, Zhang F, Ren H, Zhang Y. Analysis of Microplastics in Human Feces Reveals a Correlation between Fecal Microplastics and Inflammatory Bowel Disease Status. Environ Sci Technol. 2022 Jan 4;56(1):414-421. doi: 10.1021/acs.est.1c03924. Epub 2021 Dec 22. PMID 34935363
- [Background] Geyer R, Jambeck JR, Law KL. Production, use, and fate of all plastics ever made. Sci Adv. 2017 Jul 19;3(7):e1700782. doi: 10.1126/sciadv.1700782. eCollection 2017 Jul. PMID 28776036
- [Background] Galloway TS, Cole M, Lewis C. Interactions of microplastic debris throughout the marine ecosystem. Nat Ecol Evol. 2017 Apr 20;1(5):116. doi: 10.1038/s41559-017-0116. PMID 28812686
- [Background] Renzi M, Blaskovic A. Litter & microplastics features in table salts from marine origin: Italian versus Croatian brands. Mar Pollut Bull. 2018 Oct;135:62-68. doi: 10.1016/j.marpolbul.2018.06.065. Epub 2018 Jul 6. PMID 30301081
- [Background] Lai H, Liu X, Qu M. Nanoplastics and Human Health: Hazard Identification and Biointerface. Nanomaterials (Basel). 2022 Apr 11;12(8):1298. doi: 10.3390/nano12081298. PMID 35458006
- [Background] Akhtar S, Pranay K, Kumari K. Personal protective equipment and micro-nano plastics: A review of an unavoidable interrelation for a global well-being hazard. Hyg Environ Health Adv. 2023 Jun;6:100055. doi: 10.1016/j.heha.2023.100055. Epub 2023 Apr 11. PMID 37102160
- [Background] Cox KD, Covernton GA, Davies HL, Dower JF, Juanes F, Dudas SE. Human Consumption of Microplastics. Environ Sci Technol. 2019 Jun 18;53(12):7068-7074. doi: 10.1021/acs.est.9b01517. Epub 2019 Jun 5. PMID 31184127
- [Background] Prata JC, da Costa JP, Lopes I, Duarte AC, Rocha-Santos T. Environmental exposure to microplastics: An overview on possible human health effects. Sci Total Environ. 2020 Feb 1;702:134455. doi: 10.1016/j.scitotenv.2019.134455. Epub 2019 Oct 4. PMID 31733547
- [Background] Di Fiore C, Ishikawa Y, Wright SL. A review on methods for extracting and quantifying microplastic in biological tissues. J Hazard Mater. 2024 Feb 15;464:132991. doi: 10.1016/j.jhazmat.2023.132991. Epub 2023 Nov 10. PMID 37979423
- [Background] Catarino AI, Thompson R, Sanderson W, Henry TB. Development and optimization of a standard method for extraction of microplastics in mussels by enzyme digestion of soft tissues. Environ Toxicol Chem. 2017 Apr;36(4):947-951. doi: 10.1002/etc.3608. Epub 2016 Oct 20. PMID 27583696